CLINICAL TRIAL: NCT03009773
Title: The Multitasking Rehabilitation She Enhanced Walking Speed Compared to the Simple Post Stroke Rehabilitation Task (AVC)?
Acronym: SYNCOMOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: CENTRE DE REEDUCATION FONCTIONNELLE L'ESPOIR LILLE (Unknown); CENTRE DE REEDUCATION FONCTIONNELLE SAINT-LAZARE (Unknown); Centre Régional de Médecine Physique et de Réadaptation - Les herbiers (Unknown); Centre Hospitalier Arras (Other); CH COMPIEGNE (Unknown); CH CORBIE (Unknown); CH Le Havre (Unknown); University Hospital, Lille (Other); Clinique de rééducation fonctionnelle Le Belloy (Unknown); Fondation Hopale (Unknown); Institut Médical de Breteuil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2016_843_0007
Record Dates: First submitted 2016-11-14; First posted 2017-01-04 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Subacute Stroke
Keywords: subacute stroke; multitasking rehabilitation; walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multitasking walking (Experimental): Multitasking Group: rehabilitation multitasking walking.
  Interventions: Other: rehabilitation multitasking walking.
- walking simple task (Active Comparator): Simple task group : Traditional walking rehabilitation
  Interventions: Other: Traditional walking rehabilitation

INTERVENTIONS:
Other: rehabilitation multitasking walking. — rehabilitation multitasking walking.
  Arms: multitasking walking
Other: Traditional walking rehabilitation — Traditional walking rehabilitation
  Arms: walking simple task

SUMMARY:
Stroke is the leading cause of severe disability in adults. The first cause of alterations in the quality of life and autonomy in these patients are disorders of walking and the balance. They are the leading cause of falls responsible for important medical, surgical and economic complications as well as a reactionary social isolation.

The techniques of rehabilitation of walking to the subacute phase of a stroke are usually based on automatic walking.Off walking is a complex activity usually performed in everyday life in association with multiple tasks. It is therefore interesting to re-educate walking in dual task or even in multitasking.

ELIGIBILITY:
Inclusion Criteria:

* Major: age between 18 and 90 years
* Hospitalized for ischemic or hemorrhagic hemispheric stroke confirmed by CT or MRI <6months
* walking disorder with the possibility of walking 10 meters with or without technical assistance (speed <1.2m / s)
* verbal understanding with complex orders
* Affiliates to social security

Exclusion Criteria:

* Brainstem stroke or cerebellar
* Hypoacusia annoying understanding
* Visual gene embarrassing awarding
* severe aphasia: no understanding of complex orders
* neurological or musculoskeletal history affecting walking
* Participation in interventional research protocol in motor rehabilitation of the lower limb or cognitive
* Patient under guardianship or deprived of liberty
* pregnant women, parturient women or lactating (art L.1121-5)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Measure walking speed | 6 months
  Speed of the simple task of walking 10 meters testing.

SECONDARY OUTCOMES:
Description of different types of walking disorders and balance in the subacute phase of stroke | inclusion
  Currently no clinical scale exists in the literature at our knowledge. The walk of the patients will be qualitatively analyzed by the investigator in order to measure the prevalence of the different clinical categories of walking disorders according to their semiological characteristics
Score neuromotor the lower limb | 6 months
  Score neuromotor the lower limb: Fugl Meyer
Dynamic equilibrium to TUG single and double cognitive task | 6 months
  Dynamic equilibrium to TUG single and double cognitive task
Walking speed double cognitive task | 6 months
  Walking speed double cognitive task
Executive functions: a battery of neuropsychological | 6 months
  Executive functions: a battery of neuropsychological
Autonomy: FUNCTIONAL INDEPENDENCE MEASUREMENT | 6 months
  Autonomy: FUNCTIONAL INDEPENDENCE MEASUREMENT
EVA Quality of life | 6 months
  EVA (Visual Analogic Scale) quality of life
Correlation of cognitive gains with the gain of the walking speed of 10 meters | 6 months
  Correlation of cognitive gains with the gain of the walking speed of 10 meters
anatomoclinical correlations | 6 months
  Lesion score of gray matter and white matter (Volumetry on sequences 3DT1 and Flair) Cerebral

CONTACTS AND LOCATIONS:
Overall Officials: Sophie TASSEEL-PONCHE, Doctor, Study Director — CHU Amiens-Picardie France; Eric VERIN, professor, Principal Investigator — University Hospital, Rouen; Etienne ALLART, Doctor, Principal Investigator — CHRU de Lille; DEMAILLE Samantha, professor, Principal Investigator — CRF 4Espoir Lille; Valérie LECLERCQ-DONTGEZ, Doctor, Principal Investigator — Les 3 vallées; Haykal ELLEUCH, Doctor, Principal Investigator — CH Arras; Marie DECOCQ-DEMICHEL, Doctor, Principal Investigator — CH Le Belloy; Pascal RIGAUX, Doctor, Principal Investigator — CH Berck Sur Mer; Sabine POL-ROUX, Doctor, Principal Investigator — CH Compiègne; Sofiane LARIBI, Doctor, Principal Investigator — CH Breteuil; Skander MOALLA, Doctor, Principal Investigator — Centre Hospitalier de Beauvais
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Derived] Tasseel-Ponche S, Roussel M, Toba MN, Sader T, Barbier V, Delafontaine A, Meynier J, Picard C, Constans JM, Schnitzler A, Godefroy O, Yelnik AP. Dual-task versus single-task gait rehabilitation after stroke: the protocol of the cognitive-motor synergy multicenter, randomized, controlled superiority trial (SYNCOMOT). Trials. 2023 Mar 8;24(1):172. doi: 10.1186/s13063-023-07138-x. PMID 36890548